CLINICAL TRIAL: NCT06454903
Title: Developing a Smartphone Application to Support the Functional Needs of Veterans in Medication Treatment for Opioid Use Disorder
Brief Title: Developing a Smartphone Application to Support Veteran Opioid Use Disorder Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D5015-W; IK2RX005015-01A1 (NIH)
Record Dates: First submitted 2024-05-29; First posted 2024-06-12 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Opioid-Related Disorders; Psychosocial Functioning; Quality of Life
Keywords: Opioid-Related Disorders; Psychosocial Functioning; Quality of Life; Mobile Applications; Smartphone Apps; Acceptance and Commitment Therapy; User-Centered Design
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Stages 1 of this project will focus on developing content for a smartphone intervention (ACT to RECOVER) with input from stakeholders; Stage 2 will conduct iterative usability assessment of a beta version of ACT to RECOVER to via iterative small waves of field-testing to assess content acceptability and system usability; Stage 3 will conduct a Phase 1b randomized clinical trial, examining the acceptability and feasibility of comparing ACT to RECOVER to a smartphone-based symptom monitoring control group. Outcomes within Stage 3 will include treatment acceptability, procedural feasibility, and assessment of changes in psychosocial functioning and symptoms of opioid use disorder.
Who Masked: Outcomes Assessor
Masking Description: Study investigators will not inform outcome assessors during Stage 3 (Phase 1b clinical trial) of participant condition assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): This Phase 3 (Stage 1b RCT) Arm will consist of n = 20 Veterans (anticipated enrollment) who will receive the prototype ACT to RECOVER smartphone intervention for 4 weeks.
  Interventions: Behavioral: ACT to RECOVER
- Control (Sham Comparator): This Phase 3 (Stage 1b RCT) Arm will consist of n = 20 Veterans (anticipated enrollment) who will be assigned to receive a smartphone-based symptom-monitoring program for 4 weeks.
  Interventions: Behavioral: Smartphone-based Symptom-Monitoring

INTERVENTIONS:
Behavioral: ACT to RECOVER — During Phase 3 (Stage 1b RCT), the treatment condition will employ ACT to RECOVER. ACT to RECOVER will be a smartphone app designed to act as a flexible, semi-structured, user-friendly adjunct to standard medication treatment for opioid use disorder. Content will include components appropriate for either self-management and/or use with providers. ACT to RECOVER will be designed to have major ACT-focused modules completable within 1 month.
  Other Names: Treatment
  Arms: Treatment
Behavioral: Smartphone-based Symptom-Monitoring — During Phase 3 (Stage 1b RCT), the control condition will employ a smartphone-based symptom monitoring program in an effort to provide a balanced alternative to the treatment condition with respect to attention, time using a mobile application, and nonspecific intervention effects. This condition will not, however, include any content or components from the Prototype Digital Intervention hypothesized to produce active clinical effects.
  Other Names: Control
  Arms: Control

SUMMARY:
Opioid Use Disorder (OUD) is a complex, chronic condition affecting nearly 70,000 Veterans who can experience significantly reduced quality of life (e.g., poorer social, occupational, and health-related functioning). VA clinics providing Medication treatment for OUD (MOUD; e.g., buprenorphine, methadone), the 1st-line treatment for OUD, often face challenges in also attempting to treat Veteran functional needs, which may require them to extend beyond their available resources to provide support. There is an urgent need for functionally impactful and accessible treatments for Veterans in MOUD.

Acceptance and Commitment Therapy (ACT) is a well-suited framework to support the functioning of Veterans in MOUD with over 20 years of research support. However, the traditional practice ACT requires a trained clinician to provide weekly, hour-long therapy sessions (typically for 12-16 weeks) and may be too burdensome for MOUD clinics to use alongside standard care.

Fortunately, emerging research suggests that mobile health interventions (MHIs; e.g., smartphone apps) can overcome many of these pragmatic barriers. MHIs can efficiently deliver functionally-focused treatments focused on Veteran functioning in "real-world" settings, through minimally burdensome and accessible formats. Currently however, no MHI's targeting functioning exist for Veterans in MOUD.

The proposed study will address this gap by developing and evaluating an early prototype of a targeted smartphone app designed to enhance the functional outcomes of Veterans receiving MOUD called "ACT to RECOVER" (Acceptance and Commitment Therapy to Reach Empowerment through Commitment, Openness, and Valuing Experiences in Recovery).

The study will occur in 3 phases:

Phase 1: Development. Develop content for ACT to RECOVER using Veteran (n=10) and provider feedback (n=10).

Phase 2: Iterative Usability Assessment. Conduct field testing (3 rounds, n=4-5 per round) to refine ACT to RECOVER format, acceptability, and usability.

Phase 3: Pilot ACT to RECOVER in a Stage 1b Randomized Controlled Trial (RCT). Conduct a pilot trial to compare ACT to RECOVER (n=20) to a smartphone-based symptom monitoring control group (n=20).

* (3a) Evaluate the acceptability and feasibility of each condition's app and study procedures.
* (3b) Explore changes in functional (e.g., values-based living, quality of life) and clinical outcomes (e.g., illicit opioid use) which will be key outcomes in future efficacy testing.

DETAILED DESCRIPTION:
PHASE 1: Initial Development of the ACT to RECOVER System Phase 1: Development Phase (Months 0-15; 15 months): Veterans in MOUD (n=10) and VA MOUD clinical staff (n=10) will provide feedback and input on the intervention content drafts developed by the study team.

ACT to RECOVER Content. ACT to RECOVER will be designed to act as a flexible, semi- structured, user-friendly mobile application adjunct to MOUD. Content will include components appropriate for either self-management and/or use with providers. ACT to RECOVER will be designed to have major ACT-focused modules completable within 1 month, though Veterans will be able to continue using the app and its features after study completion, upon request. Core content for ACT to RECOVER's modules will be adapted from major ACT texts (e.g., Hayes and colleagues' Acceptance and Commitment Therapy: The Process and Practice of Mindful Change) and technology (e.g., VA ACT Coach). Core Content modules will cover: 1) Behavior change and addiction triggers, 2) values clarification, 3) acceptance, 4) cognitive defusing, 5) committed action, and 6) willingness. Additional "general" content modules will also be included (e.g., providing support for medication and appointment tracking) to support treatment engagement.

Phase 1 Qualitative Interviews Interview Guide. Interviews will include open-ended questions on ACT to RECOVER's acceptability, feasibility of engagement, potential concerns, and initial reactions. Interview questions are based on the Practical, Robust Implementation and Sustainability Model (PRISM).

Interview Analysis Qualitative data analysis will use a thematic approach with the goal of ascertaining intervention acceptability, feasibility of engagement, and referral issues. Two independent reviewers will code each interview transcription using open-ended coding. Each element will be summarized separately, and themes and key points will be generated to assess data saturation. Two reviewers will analyze the qualitative data using modified grounded coding to identify themes from audio recordings after each interview. Intervention areas will be modified as feedback is given. Each set of interviews will take place with 3-4 participants per group. The number of changes needed for each intervention area will be tracked; it is anticipated that less intervention refinement will be needed by the end of the interview cycle. If later interviews still suggest a need for significant refinement (e.g., increasing number of changes needed), further testing will be done.

PHASE 2: Iterative Usability Testing Phase 2: Pilot Evaluation of Intervention Components in Field-Based Iterative Usability Testing (Months 15-33; 18 months): Veterans will be recruited in MOUD (N=12-15) to conduct usability and content acceptability testing of ACT to RECOVER across 3 iterative waves (n=4-5 per wave).

Iterative Usability Assessment Procedures Eligible Veterans will come to the VACHS West Haven campus to complete baseline measures. Following, Veterans will be provided with a smartphone containing a beta-version of ACT to RECOVER. First, Veterans will be walked through portions of the mobile application and its user interface. Different images for options of the ACT to RECOVER app, as well as a PowerPoint with information about the user interface will be shown to simulate the intervention and its user interface. Second, Veterans will be provided with written instructions and asked to do a behavioral walk-through of a portion of the ACT to RECOVER system using the beta app version and provided PowerPoint slides. Third, Veterans will be asked to move through the ACT to RECOVER system unguided. Throughout, a combined usability and contextual interview approach will be used in which participant system use is recorded while they are asked questions about their engagement and preferences. Finally, participants will complete acceptability and usability measures, as well as a semi-structured qualitative exit interview. An average of 2 weeks between waves to allow time for Geisel Software Inc. to address identified functionality and interface concerns. Go/no-go limits to determine whether Phase 3 should commence are set a priori (see section 6b. Outcome Measures).

Data Collection and Analysis Quantitative statistics will be computed and reported to describe the sample and assess for pre-defined go/no-go limits for the next Phase. In accordance with an adapted Integrated Technology Acceptance Model (ITAM) framework, correlations will also be assessed between health factors and demographic information with intrinsic motivation, perceived ease of use/usefulness, and behavioral intent to use ACT to RECOVER. It is expected that positive correlations between all ITAM constructs will be present.

Qualitative Combined Usability and Contextual Interview Analysis. During usability sessions, participants will assess ACT to RECOVER using a "think-aloud" protocol, verbalizing their thoughts as they navigate the app. After a period of exploration with the app, the research staff will use a pre-created protocol to ask Veterans to perform a series of tasks (e.g., accessing different modules). Session and on-screen recording will occur alongside real-time observation. Additionally, Veterans will complete a series of brief usability questionnaires following user testing and the qualitative interview.

A modified consensual qualitative research (CQR) approach will be used to code the session transcriptions. Research team investigators initial codebook based on key activities and questions in the user-testing protocol will be developed and employed for identifying usability themes within screen-recorded videos, with additional research staff identified to act as a code auditor: (a) Two coders utilize the initial codebook throughout data analysis to foster multiple perspectives; (b) consensus is reached between coders about the meaning of the data; (c) at least one auditor must check the work of the primary team of judges to minimize potential bias; and (d) domain and theme frequency are reported.

Themes will then be categorized according to the following CQR groupings: general (include all or all but one of the cases), typical (include more than half of the cases up to the cut off for general), and variant (at least two cases up to the cutoff for typical). General comments will be classified regarding usability as necessary to include in iterative development, typical and variant will be discussed within the research group to decide upon potential ways to incorporate this feedback into intervention refinement. Feedback will then be triangulated per testing wave by 1) summarizing suggested changes, 2) obtaining study team input, and 3) meeting with the software development team to implement changes.

PHASE 3: Stage 1b Pilot RCT Phase 3: Stage 1b Pilot RCT (Months 33-60; 27 months): A Stage 1b RCT pilot will be conducted to assess the acceptability (treatment satisfaction, perceived ease of use and usefulness, behavioral intent to use, actual use) and feasibility (recruitment, treatment receptivity, sustained participation, and attrition in each condition) of comparing ACT to RECOVER (n=20) to a smartphone-based symptom monitoring control condition (n=20). Phase 3 will focus on (3a) assessing the acceptability and feasibility of the intervention and research procedures and (3b) exploring the data characteristics of, and describing changes in, functional (e.g., values-consistent living) and clinical outcomes (e.g., illicit opioid use).

Stage 1b Pilot RCT Procedures At the start of this visit, research staff will confirm participant eligibility and verify informed consent. Following, Veterans will complete baseline demographic and health measures, as well as relevant outcome measures. Veterans will have been randomized to receive either ACT to RECOVER (treatment arm) or smartphone-based symptom monitoring (control) condition prior to their baseline study visit, with instructions for the appropriate app download and use provided during the baseline session (please refer to section 7. Arms & Interventions for details). Veterans will be asked to use the respective condition's app over the next 5 weeks and to attend midpoint (week 2), endpoint (week 4), and follow-up (week 5) study visits, during which indicated measures will be collected (see section 6b. Outcome Measures).

Semi-structured qualitative exit interview. A 30-minute, semi-structured qualitative interview will be conducted with Veterans in both arms during the endpoint assessment, to further assess acceptability, feasibility, usability, and dissemination issues. Questions will inquire about any problems with app access and use, perceived effects, if Veterans would recommend the app to a friend, and recommended changes.

Data Management and Statistical Analysis Power analysis. Consistent with the NIH Stage model for intervention development, this Stage 1b RCT will focus on determining the acceptability and feasibility of a given intervention and study procedures (vs. efficacy testing), and accordingly proposes a sample of N=40 (n=20 eligible participants per group).

Primary Analyses and Hypotheses, Stage 1b RCT - Aim 3a: Acceptability and feasibility of study intervention and procedures. Targets for aim 3a include descriptively assessing if the ACT to RECOVER and smartphone-based symptom monitoring control apps reach thresholds for intervention acceptability, feasibility, and maintenance of usability thresholds (see section 6b Study Outcomes for details on these measures and thresholds). If study thresholds are not met, the study team and Geisel Software's development team will convene to discuss further intervention and/or study procedure refinement, which may include additional data collection until thresholds are met. Threshold achievement would indicate the ACT to RECOVER system and trial procedures are suitable for a subsequent efficacy trial.

Aim 3a Hypotheses:

It is hypothesized that all constructs will positively correlate with each other (e.g., greater medical care satisfaction, info seeking, and health care need will positively correlate with intrinsic motivation for app use, which will positively correlate with perceived ease of use and usefulness, behavioral intention to use the app, and ultimately with actual app use). Analysis of post-intervention interviews will also be done using notes taken by study staff during the exit interview; interviews will also be audiotaped and transcribed for later analysis. Research staff will apply CRQ qualitative analytic techniques to these data (e.g., coding and extracting major themes) to assess barriers and facilitators to app use per condition.

Secondary Analyses, Stage 1b RCT - Aim 3b: Descriptive analyses to provide preliminary empirical evidence for a subsequent efficacy trial and inform its design.

Consistent with the Stage of Phase 3's proposed trial, Aim 3b will also assess if the proposed study procedures are suitable to collect the requisite data for future efficacy testing. For each condition, the study team will calculate descriptive statistics, assess univariate distributions, explore bivariate relationships, and conduct paired-samples t-tests to evaluate the potential changes in functional and clinical outcomes within-subjects. These analyses will examine baseline in comparison to each subsequent study interval (i.e., baseline vs. midpoint, baseline vs. endpoint, baseline vs. 5-week follow-up), and will be conducted on the whole sample, as well as stratified by group.

Aim 3b Hypotheses:

It is hypothesized that those in the ACT to RECOVER condition will demonstrate an increase in values-based living, quality of life, and MOUD compliance for Veterans in the ACT to RECOVER condition, as well as a decrease in behavioral avoidance, illicit opioid use, and substance-related problems.

ELIGIBILITY:
Inclusion Criteria:

For the Phase 3, Stage 1b RCT we will be recruiting Veterans enrolled within the VA CT Healthcare System with:

* Current diagnosis of Opioid Use Disorder (OUD) indicated by either DSM-5-TR or ICD-9 or -10 codes
* Active Medication treatment for OUD prescription for buprenorphine or methadone (in any formulation)
* A working smartphone with wireless capabilities (to allow for download of ACT to RECOVER) or is willing to use a study-provided smartphone
* Competency to provide written informed consent
* 18 years of age or older

Exclusion Criteria:

Participants may not:

* Have been on MOUD, in their current treatment episode (i.e., since their most recent induction), for longer than 12 consecutive months prior to their baseline visit
* Have untreated major psychiatric disorders (e.g., bipolar disorders, psychotic disorders)
* Be expressing current, active suicidal/homicidal ideation (i.e., current intent to harm themselves or someone else)
* Have any cognitive/medical impairment precluding study participation or use of smartphones/smartphone applications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Theoretical Framework of Acceptability (TFA) scale | Phase 3 (Stage 1b RCT): Baseline (week 0); Endpoint (Week 4)
  The Theoretical Framework of Acceptability provides a rigorous framework for assessing the acceptability of health information technology, offering both prospective and retrospective acceptability scales, which respectively assess how acceptable one believes they will find a health intervention and how acceptable they found the intervention after use. We will use the prospective scale (i.e., assessing how acceptable participants think the ACT to RECOVER app would be if they were to use as part of their treatment). The TFA's scale asks participants to rate 7 dimensions of acceptability (affective attitude towards a health intervention, burden, value alignment, understanding of intervention functioning, perceived benefit, perceived effectiveness, and self-efficacy) on a 5-point scale, with avg.'s >3 indicating minimum degrees of acceptability.
App usage: Openings | Phase 3 (Stage 1b RCT): Tracked continuously from Baseline (week 0) through Follow-up (week 5)
  Continuously-recorded via smartphone apps in respective conditions as a frequency count of the number of times a respective app is opened.
App usage: Duration | Phase 3 (Stage 1b RCT): Tracked continuously from Baseline (week 0) through Follow-up (week 5)
  Continuously-recorded via smartphone apps in respective conditions as the total duration of time (as number of minutes) spent using the respective app.
Enrollment: Enrollment Rate | End of Month 60 (Final month of project, upon which completion of Phase 3 (Stage 1b RCT) recruitment and follow-up is anticipated to complete)
  Participant enrollment rate. Study target is >2 participants/month on avg., assessed upon completion of Stage 3 study procedures.
App usage: Completion | Phase 3 (Stage 1b RCT): Tracked continuously from Baseline (week 0) through Follow-up (week 5)
  Continuously-recorded via smartphone apps in respective conditions as the number of module/symptom reports completed. Targets are for an avg. of >3/6 ACT to RECOVER modules + 1 General module completed (ACT to RECOVER condition) or an avg. of >15/30 days of symptom monitoring reports (symptom monitoring control condition).
Enrollment: Attrition | End of Month 60 (Final month of project, upon which completion of Phase 3 (Stage 1b RCT) recruitment and follow-up is anticipated to complete)
  Percentage of participant attrition. Study target is <35.5% per study arm, assessed upon completion of Stage 3 study procedures.
Systems Usability Scale (SUS) | Phase 3 (Stage 1b RCT): Endpoint (Week 4)
  The SUS is a 10-item measure, scored on a 5-point Likert scale from Strongly Disagree (1) to Strongly Agree (5), that assesses human-computer interaction. The SUS generates a subjective evaluation score using a globally accepted scale and to understand if the system in its current form is sufficiently usable. To calculate the SUS score, first sum the score contributions from each item. Each item's score contribution will range from 0 to 4. For items 1,3,5,7,and 9 the score contribution is the scale position minus 1. For items 2,4,6,8 and 10, the contribution is 5 minus the scale position. Multiply the sum of the scores by 2.5 to obtain the overall value of system usability. SUS scores have a range of 0 to 100, with higher scores suggesting greater system usability. A SUS score above 68 (study target) is regarded as above average, and a SUS score above 80 is regarded as high and a score above which participants are likely to recommend the product to friends.

SECONDARY OUTCOMES:
Usability Survey | Phase 3 (Stage 1b RCT): Endpoint (Week 4)
  The usability survey items are drawn from a questionnaire developed by Wilson and Lankton (2004) to measure a range of health information technology areas. Each item is scored on a 7 point Likert scale where 1 = strongly disagree and 7 = strongly agree. There are 8 subscales: 1. Satisfaction with Medical Care Scale (3 items, range 3 - 21); 2. Health Knowledge Scale (2 items, range 2 to 14); 3. Internet Dependence Scale (4 items, range 4 to 28); 4. Information-seeking Preference Scale (4 items, range 4 to 28); 5. Intrinsic Motivation Scale (3 items, range 3 to 21); 6. Perceived Ease of Use Scale (3 items, range 3 to 21); 7. Perceived Usefulness: Extrinsic Motivation Scale (3 items, range 3 to 21); 8. Behavioral Intention to Use E-health Scale (2 items, range 2 - 14). For each scale, items are summed, with higher score indicating greater levels of satisfaction, knowledge, dependence, information preference, motivation, ease of use, usefulness, and intention to use the system.
Values-based living (VQ) | Phase 3 (Stage 1b RCT): Baseline (Week 0); Midpoint (Week 2); Endpoint (Week 4); Follow-up (Week 5)
  Valued living will be assessed using the Valuing Questionnaire (VQ), which assesses the extent to which personal values have been enacted within the past week. It is designed to capture the quality of valued action (i.e., the extent to which behaviors accord with what one values) using everyday language and without reference to specific life domains.
Multidimensional Experiential Avoidance Questionnaire (MEAQ | Phase 3 (Stage 1b RCT): Baseline (Week 0); Midpoint (Week 2); Endpoint (Week 4); Follow-up (Week 5)
  A 62-item self-report measure of experiential avoidance, including subscales on Behavioral Avoidance (11 items, range 11 to 66), Distress Aversion (13 items, range 13 to 78), Procrastination (7 items, range 7 to 42), Distraction & Suppression (7 items, range 7 to 42), Repression & Denial (13 items, range 13 to 78), and Distress Endurance (11 items, range 11 to 66). The scale for all items ranges from 1 (strong disagree) to 6 (strongly agree). Greater scores within each subscale indicate greater levels of the named construct. A total score can be obtained with the following calculation: Behavioral Avoidance + Distress Aversion + Procrastination + Distraction & Suppression + Repression & Denial + (77 - Distress Endurance).
Veteran's RAND 36 (VR-36) | Phase 3 (Stage 1b RCT): Baseline (Week 0); Midpoint (Week 2); Endpoint (Week 4); Follow-up (Week 5)
  Quality of Life will be assessed using the Veteran's RAND 36-item Health Survey (VR-36), which is designed to assess health-related quality of life with respect to role limitations, social and physical functioning, general and mental health, energy and fatigue, and bodily pain. It is often summarized into physical and mental functioning components, and is one of the most widely utilized and valid measures of physical and psychological well-being.
Timeline Follow Back for Illicit Opioid Use and Medication Compliance | Phase 3 (Stage 1b RCT): Baseline (Week 0); Midpoint (Week 2); Endpoint (Week 4); Follow-up (Week 5)
  Illicit opioid use and compliance with medication treatment regiments for opioid use disorder will be assessed using Timeline Followback procedures (TLFB) outlined by McCann et al. (2024) for opioid use disorder. These assessments will produce a count of days of illicit opioid and MOUD use during the past month (at baseline) and since the prior assessment timepoint (at midpoint, endpoint, and 5-week follow-up).
Short Inventory of Problems - Revised (SIP-R) | Phase 3 (Stage 1b RCT): Baseline (Week 0); Midpoint (Week 2); Endpoint (Week 4); Follow-up (Week 5)
  The SIP-R will provide a self-report assessment of the adverse consequences of substance use. The SIP-R asks participants to indicate the frequency of 17 different substance-related consequences, which are scored from 0-3. Item responses are then summed to produce a total score, as well as five subscales (physical, social, intrapersonal, interpersonal, and impulse control). Higher scores are indicative of greater substance-related problems and poorer treatment engagement (Kiluk et al., 2013).
Usability Survey: Perceived Usefulness: Extrinsic Motivation Scale | Phase 3 (Stage 1b RCT): Endpoint (Week 4)
  The Perceived Usefulness: Extrinsic Motivation Scale consists of 3 items drawn from Wilson and Lankton (2004) Usability Survey. Each item is scored on a 7-point Likert scale where 1 = strongly disagree and 7 = strongly agree. Scale items are summed, with higher score indicating greater belief that using and interacting with a given health intervention will be beneficial to one's healthcare.
Usability Survey: Behavioral Intention to Use E-health Scale | Phase 3 (Stage 1b RCT): Endpoint (Week 4)
  The Behavioral Intention to Use E-health Scale consists of 2 items drawn from Wilson and Lankton (2004) Usability Survey. Each item is scored on a 7-point Likert scale where 1 = strongly disagree and 7 = strongly agree. Scale items are summed, with higher score indicating greater intent to use a given health intervention.
Values-based living (VQ): Values Progress | Stage 3 Phase 1b RCT: Baseline (Week 0); Midpoint (Week 2); Endpoint (Week 4); Follow-up (Week 5)
  Progress towards one's values will be assessed using the Valuing Questionnaire's (VQ's) Values Progress subscale, which assesses the extent to which personal values have been enacted within the past week. It is designed to capture the quality of valued action (i.e., the extent to which behaviors accord with what one values; e.g., "I made progress in the areas of my life I care most about") and contains items 3, 4, 5, 7, and 9 from the VQ. Subscale items are scored on a 0-6 Likert scale (0 = Not at all true, 6 = Completely true) and are summed with higher scores indicating greater values progress.
Values-based living (VQ): Values Obstruction | Stage 3 Phase 1b RCT: Baseline (Week 0); Midpoint (Week 2); Endpoint (Week 4); Follow-up (Week 5)
  Obstruction of values will be assessed using the Valuing Questionnaire's (VQ's) Values Obstruction subscale, which assesses the extent to which one feels they have been prevented from acting in-concert with personal values within the past week (e.g., "Difficult thoughts, feelings, or memories got in the way of what I really wanted to do") and contains items 1, 2, 6, 8, and 10 from the VQ. Subscale items are scored on a 0-6 Likert scale (0 = Not at all true, 6 = Completely true) and are summed with higher scores indicating greater values obstruction.
Multidimensional Experiential Avoidance Questionnaire (MEAQ) | Stage 3 Phase 1b RCT: Baseline (Week 0); Midpoint (Week 2); Endpoint (Week 4); Follow-up (Week 5)
  A 62-item self-report measure of experiential avoidance, including subscales on Behavioral Avoidance (11 items, range 11 to 66), Distress Aversion (13 items, range 13 to 78), Procrastination (7 items, range 7 to 42), Distraction & Suppression (7 items, range 7 to 42), Repression & Denial (13 items, range 13 to 78), and Distress Endurance (11 items, range 11 to 66). The scale for all items ranges from 1 (strong disagree) to 6 (strongly agree). Greater scores within each subscale indicate greater levels of the named construct. A total score can be obtained with the following calculation: Behavioral Avoidance + Distress Aversion + Procrastination + Distraction & Suppression + Repression & Denial + (77 - Distress Endurance).
Veteran's RAND 36 (VR-36): Physical Component Score | Phase 3 Stage 1b RCT: Baseline (Week 0); Midpoint (Week 2); Endpoint (Week 4); Follow-up (Week 5)
  Quality of Life will be assessed using the Veteran's RAND 36-item Health Survey (VR-36), which is designed to assess health-related quality of life with respect to role limitations, social and physical functioning, general and mental health, energy and fatigue, and bodily pain. Computer-based algorithms can be used to calculate physical and mental functioning component scores. The Physical Component Score (PCS) provides a greater emphasis on questions of general health, physical functioning, role enactment, and bodily pain.
Veteran's RAND 36 (VR-36): Mental Health Component Score | Phase 3 Stage 1b RCT: Baseline (Week 0); Midpoint (Week 2); Endpoint (Week 4); Follow-up (Week 5)
  Quality of Life will be assessed using the Veteran's RAND 36-item Health Survey (VR-36), which is designed to assess health-related quality of life with respect to role limitations, social and physical functioning, general and mental health, energy and fatigue, and bodily pain. Computer-based algorithms can be used to calculate physical and mental functioning component scores. The Mental health Component Score (PCS) provides a greater emphasis on questions of emotional well-being, mental health and perceptions of vitality, and social functioning.
Timeline Follow Back: Illicit Opioid Use | Phase 3 Stage 1b RCT: Baseline (Week 0); Midpoint (Week 2); Endpoint (Week 4); Follow-up (Week 5)
  Illicit opioid use opioid use will be assessed using Timeline Followback procedures (TLFB) outlined by McCann et al. (2024) for opioid use disorder. These assessments will produce a count of days of illicit opioid use during the past month (at baseline) and since the prior assessment timepoint (at midpoint, endpoint, and 5-week follow-up).
Timeline Follow Back: Medication Compliance | Phase 3 Stage 1b RCT: Baseline (Week 0); Midpoint (Week 2); Endpoint (Week 4); Follow-up (Week 5)
  Compliance with medication treatment regiments for opioid use disorder will be assessed using Timeline Followback procedures (TLFB) outlined by McCann et al. (2024) for opioid use disorder. These assessments will produce a count of days of MOUD use during the past month (at baseline) and since the prior assessment timepoint (at midpoint, endpoint, and 5-week follow-up).
Short Inventory of Problems - Revised (SIP-R) | Stage 3 Phase 1b RCT: Baseline (Week 0); Midpoint (Week 2); Endpoint (Week 4); Follow-up (Week 5)
  : The SIP-R will provide a self-report assessment of the adverse consequences of substance use. The SIP-R asks participants to indicate the frequency of 17 different substance-related consequences, which are scored from 0-3. Item responses are then summed to produce a total score, as well as five subscales (physical, social, intrapersonal, interpersonal, and impulse control). Higher scores are indicative of greater substance-related problems and poorer treatment engagement (Kiluk et al., 2013).

CONTACTS AND LOCATIONS:
Overall Officials: Noah R Wolkowicz, PhD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (1):
- VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No